CLINICAL TRIAL: NCT06270589
Title: Supporting High-intensity Interval Training With Mindfulness for Enhancing Childhood Executive Function
Brief Title: Acute Effects of High-intensity Interval Training With Mindfulness-based Recovery on Executive Function in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: University of Oregon (Other)
Responsible Party: Principal Investigator, Shih-Chun Kao, Assistant Professor, Purdue University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2023-1684
Record Dates: First submitted 2024-01-29; First posted 2024-02-21 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers
Keywords: Interval Exercise; Mindfulness; Executive function; Brain function; Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- A Single Bout Of Mindful High-Intensity Interval Training (Mindful HIIT) (Experimental)
  Interventions: Behavioral: MF-HIIT
- A Single Bout Of High-Intensity Interval Training (HIIT) (Active Comparator)
  Interventions: Behavioral: HIIT-only
- A Single Bout Of Mindfulness (Active Comparator)
  Interventions: Behavioral: MF-only
- A Single Bout Of Sitting Rest (Other)
  Interventions: Behavioral: Sitting rest

INTERVENTIONS:
Behavioral: MF-HIIT — A single bout of 20-min MF-HIIT protocol delivered through a motor-driven treadmill. The protocol will start with a 1.5-min warm-up, then a 16.5-min main exercise (6 x 90s exercise intervals separated by 5 x 90s mindful intervals), and finally a 2-min cool-down.
  Arms: A Single Bout Of Mindful High-Intensity Interval Training (Mindful HIIT)
Behavioral: MF-only — A single bout of 20-min intervention mindfulness intervention that includes 5 x 90s mindful intervals separated by sitting rest
  Arms: A Single Bout Of Mindfulness
Behavioral: HIIT-only — A single bout of 20-min HIIT protocol delivered through a motor-driven treadmill. The protocol will start with a 1.5-min warm-up, then a 16.5-min main exercise (6 x 90s exercise intervals separated by 5 x 90s rest intervals), and finally a 2-min cool-down.
  Arms: A Single Bout Of High-Intensity Interval Training (HIIT)
Behavioral: Sitting rest — Participants will sit in a comfortable chair, placed on the treadmill, while watching a HIIT video without mindfulness instructions for 20 minutes.
  Arms: A Single Bout Of Sitting Rest

SUMMARY:
The goal of this randomized cross-over trial is to learn about the effect of a single bout of 20-min mindfulness-based high-intensity interval training (MF-HIIT), MF-only, and HIIT-only in relative to sitting rest on executive function (EF) in 10-12 years old children. The main question it aims to answer are:

Question 1: Whether a single bout of 20-min MF-HIIT has larger beneficial effect on EF performance than that following a 20-min session of MF-only and HIIT-only in relative to the sitting rest

Question 2: Whether a single bout of 20-min MF-HIIT has a larger beneficial effect on brain functioning, as measured by the N2 and P3 components of event-related potential (ER) during EF performance than that following a 20-min session of MF-only and HIIT-only in relative to the sitting rest

Participants will visit the laboratory on 5 separate days (> 2-day washout between days) in which they have not previously participated in structured physical activities.

Participants will complete the testing and/or receive treatments below:

Day 1:

* Kaufman Brief Intelligence Test (KBIT) to assess intelligence quotient
* Treadmill-based exercise test to measure cardiorespiratory fitness (maximum oxygen consumption)

Days 2-5

* Each day, participants will complete each of the four intervention conditions (MF-HIIT, MF-only, HIIT-only, sitting)
* Participants' heart rate and self-reported affect and rating of physical exertion will be measured
* Participants will complete a modified flanker task and a task-switching task to assess inhibitory control and cognitive flexibility
* Participants will wear an EEG cap to measure the N2 and P3 components of the event-related potential during the inhibitory control and cognitive flexibility performance

Researcher will compare the cognitive outcome measures following the MF-HIIT, MF-only, and HIIT-only conditions with the sitting condition to see if MF and HIIT has beneficial effects on children's EF.

Further, researcher will compare the cognitive outcome measures following the MF-HIIT compared with MF-only and HIIT-only conditions to see if combining MF with HIIT has greater beneficial effects on children's EF than MF and HIIT alone.

ELIGIBILITY:
Inclusion Criteria:

* Age between 10-12 years old
* Intelligence Quotient ≥ 85
* Capable of performing exercise based on pre-participation health screening
* No formal diagnosis of cognitive disorders (e.g., attention deficit hyperactivity disorder) and neurological diseases (e.g., epilepsy)

Exclusion Criteria:

* Age outside of the range of 10-12 years old
* Intelligence Quotient < 85
* No capable of performing exercise based on pre-participation health screening
* Has formal diagnosis of cognitive disorders (e.g., attention deficit hyperactivity disorder) and neurological diseases (e.g., epilepsy)

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Inhibition speed | At the baseline before and about 10-min after the 20-min intervention on Day 2, Day 3, Day 4, and Day 5.
  Inhibition speed will be assessed by the response time (ms) during a child-friendly flanker task.
Inhibition accuracy | At the baseline before and about 10-min after the 20-min intervention on Day 2, Day 3, Day 4, and Day 5.
  Inhibition accuracy will be assessed by the response accuracy (%) during a child-friendly flanker task.
Shifting speed | At the baseline before and about 10-min after the 20-min intervention on Day 2, Day 3, Day 4, and Day 5.
  The shifting speed will be assessed by the response time (ms) during a child-friendly switching task.
Shifting accuracy | At the baseline before and about 10-min after the 20-min intervention on Day 2, Day 3, Day 4, and Day 5.
  The shifting accuracy will be assessed by the response accuracy (%) during a child-friendly switching task.
N2-ERP | At the baseline before and about 10-min after the 20-min intervention on Day 2, Day 3, Day 4, and Day 5.
  The N2 component of event-related brain potentials is a neuroelectric index of conflict processing. Increased amplitude of N2 reflects increased neural activation to detect and resolve conflicts.
P3-ERP | At the baseline before and about 10-min after the 20-min intervention on Day 2, Day 3, Day 4, and Day 5.
  The P3 component of event-related brain potentials is a neuroelectric index of attention. Increased amplitude of P3 reflects greater allocation of attentional resources and the decreased latency of P3 reflects the faster information processing speed.

SECONDARY OUTCOMES:
State Mindfulness Scale for Physical Activity (SMSPA) | Immediately after completing the 20-min intervention on Day 2, Day 3, Day 4, and Day 5.
  A developmentally-appropriate and validated 12-item, 5-point Likert scaled (0-4), instrument to measure self-reported mindfulness state in children aged above 10 years old. This measure will serve as a manipulation check on mindfulness induction during each of the 4 intervention conditions.
Rating of perceived exertion | Measure at 0 second, 90 seconds, 180 seconds, 270 seconds, 360 seconds, 450 seconds, 540 seconds, 630 seconds, 720 seconds, 810 seconds, 900 seconds, 990 seconds, 1080 seconds and 1200 seconds of the 20-min intervention on Day 2, Day 3, Day 4, and Day 5.
  The 10-point Children's OMNI rating of perceived exertion will be used as a manipulation check on the intensity of prescribed exercise for the school-based programs as well as the laboratory-based acute interventions.
Heart Rate | Heart rate will be measured at every minute (minutes 0, 1, 2, 3, 4, ...., 18, 19, 20) during the 20-min intervention on Day 2, Day 3, Day 4, and Day 5.
  Heart rate will serve as a manipulation check on the intensity of prescribed exercise.

OTHER OUTCOMES:
Dispositional mindfulness | At baseline on Day 1 before receiving any intervention
  Child and Adolescent Mindfulness Measure (CAMM) provides a validated and reliable measure of dispositional mindfulness in children using 10 items and 5-point Likert scale (0-4), with a higher total score indicating the participant is more mindful. This measure will be used as the secondary outcome measure to to check the intervention manipulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Lambert, 800 West Stadium Avenue, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No